CLINICAL TRIAL: NCT00299312
Title: Rett Syndrome Natural History: Genetic and Physical Characteristics of Rett Syndrome
Brief Title: Genetic and Physical Characteristics of Rett Syndrome
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); Greenwood Genetic Center (Other); Baylor College of Medicine (Other); Boston Children's Hospital (Other); University of Rochester (Other); Children's Hospital of Philadelphia (Other); University of Colorado, Denver (Other); Rush University Medical Center (Other); UCSF Benioff Children's Hospital Oakland (Other); University of California, San Diego (Other); Vanderbilt University (Other); University of South Florida (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Alan Percy, Professor, Pediatrics, Neurolgy, Neurobiology, Genetics, University of Alabama at Birmingham
Other Study IDs: RDCRN 5201; U54HD061222 (NIH); ARP 5201
Record Dates: First submitted 2006-03-03; First posted 2006-03-06 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Rett Syndrome; MECP2 Duplication Disorder; Rett-related Disorder
Keywords: Loss of Purposeful Hand Use Syndrome; Loss of Communication; Stereotypic Hand Movements; MECP2 mutation; MECP2 duplication; CDKL5 mutation; FOXG1 mutation
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Rett Syndrome (RTT) is a genetic brain disorder that occurs almost exclusively in females and is usually caused by a change (mutation) in the gene MECP2. The disorder is characterized by multiple developmental problems, as well as behavioral features, such as repetitive stereotypic hand movements, including hand washing, wringing, and tapping. While there is no cure for RTT, recent advances in the understanding of the disease suggest that the development of new, effective therapies is promising. This study will gather information on the genetic defects that cause RTT, the physical expressions of these defects, and disease progression. In turn, this may direct the development of future treatments. Expanded studies include individuals with MECP2 Duplication disorder, and RTT-related disorders including individuals with MECP2 mutations, but not meeting obligatory criteria for the diagnosis of RTT and individuals with mutations in CDKL5 and FOXG1 some of whom meet criteria for atypical RTT.

DETAILED DESCRIPTION:
RTT is a brain disorder that causes problems with childhood development. It is usually caused by an abnormality (mutation) in the gene MECP2. RTT can cause severe impairments in movement and communication skills, including speech and social interaction. The first signs of RTT include loss of acquired speech and loss of purposeful hand use for activities such as eating or playing. Individuals may also develop abnormal walking, repetitive hand movements, such as clapping or wringing, and abnormal breathing while awake.

Effective treatments for RTT are currently lacking. There is also inadequate information about the link between RTT clinical features and its genetic basis. In order to prepare for future clinical trials that may lead to effective therapies, it is important to collect accurate information about the characteristics of RTT and the pattern of disease progression. This study will gather historical and physical examination data to establish phenotype-genotype correlations. Data on survival and quality of life in females with RTT and males with MECP2 gene mutations will also be evaluated.

MECP2 Duplication disorder affects principally males who have one and rarely more than one additional copy of MECP2 as well as a variable number of other duplicated genes. These males have absent spoken language, shuffling gait, epilepsy, and, in some, frequent upper respiratory infections or sinusitis. Mother of these males are generally normal due to favorable skewing of X-chromosome inactivation, but in some instances may have neurodevelop-mental delays. Effective treatments are lacking. It is critical to develop phenotype-genotype correlations and longitudinal natural history data to assist the conduct of clinical trials.

RTT-related disorders feature a variety of involvements either due to MECP2, CDKL5, and FOXG1 as well as other potential causes of atypical RTT. Phenotype-genotype studies and longitudinal natural history data are essential to the conduct of future clinical trials.

Participants in this observational study will be recruited from the four sites at which the study is being conducted, as well as through the Rare Disease Clinical Research Network and the International Rett Syndrome Association (IRSA). Prior to study entry, potential participants are expected to be tested for a mutation in the MECP2 gene. No treatment will be administered at any time during this study. Study visits will occur every 6 months until the child is 6 years old and once a year thereafter. At each study visit, participants will be examined to assess physical characteristics of the disorder, such as motor behavior and disease severity. Additionally, participants will complete questionnaires about medical history, contact information, and quality of life. The first visit will last approximately 1.5 hours, and every subsequent visit will last approximately 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Meets clinical criteria for classic or variant RTT or tests positive for an MECP2 gene mutation or a MECP2 duplication or a mutation in CDKL5 or FOXG1.

Exclusion Criteria:

* Unwilling or unable to travel to study sites for annual or biannual evaluations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals fulfilling consensus clinical criteria for Classic or Variant Rett Syndrome, individuals with MECP2 mutations who do not meet the clinical criteria, or individuals who have a duplication of Xq28 including the MECP2 locus or individuals who have mutations in CDKL5 or FOXG1.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2006-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Genetic and Physical Characteristics of Rett Syndrome | July 31, 2019
  The primary endpoint is to determine the variables related to clinical outcome in terms of genotype and phenotype. The variables include growth, head circumference, stereotypic movements, periodic breathing, epilepsy, scoliosis, and longevity. Summative data are provided by the Clinical Severity Scale (CSS) and the Motor Behavioral Assessment (MBA) and specific neurophysiologic and neuroimaging studies in selected participants.

SECONDARY OUTCOMES:
Genetic and Physical Characteristics of Rett syndrome | Through July 31, 2019
  The principal secondary outcome measures include quality of life assessments of the participants (CHQ) and the principal caregiver (SF-36).

OTHER OUTCOMES:
Genetic and Physical Characteristics of Rett Syndrome, MECP2 Duplication disorder, and RTT-related conditions | July 31, 2019
  No other pre-specified outcome measures are planned

CONTACTS AND LOCATIONS:
Overall Officials: Alan K Percy, MD, Principal Investigator — University of Alabama at Birmingham
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital of Oakland, Oakland, California
  - University of California San Diego, San Diego, California
  - University of Colorado Denver, Denver, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Rochester, Rochester, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Greenwood Genetic Center, Greenwood, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Laccone F, Junemann I, Whatley S, Morgan R, Butler R, Huppke P, Ravine D. Large deletions of the MECP2 gene detected by gene dosage analysis in patients with Rett syndrome. Hum Mutat. 2004 Mar;23(3):234-44. doi: 10.1002/humu.20004. PMID 14974082
- [Background] Schanen C, Houwink EJ, Dorrani N, Lane J, Everett R, Feng A, Cantor RM, Percy A. Phenotypic manifestations of MECP2 mutations in classical and atypical Rett syndrome. Am J Med Genet A. 2004 Apr 15;126A(2):129-40. doi: 10.1002/ajmg.a.20571. PMID 15057977
- [Background] Neul JL, Fang P, Barrish J, Lane J, Caeg EB, Smith EO, Zoghbi H, Percy A, Glaze DG. Specific mutations in methyl-CpG-binding protein 2 confer different severity in Rett syndrome. Neurology. 2008 Apr 15;70(16):1313-21. doi: 10.1212/01.wnl.0000291011.54508.aa. Epub 2008 Mar 12. PMID 18337588
- [Background] Bebbington A, Anderson A, Ravine D, Fyfe S, Pineda M, de Klerk N, Ben-Zeev B, Yatawara N, Percy A, Kaufmann WE, Leonard H. Investigating genotype-phenotype relationships in Rett syndrome using an international data set. Neurology. 2008 Mar 11;70(11):868-75. doi: 10.1212/01.wnl.0000304752.50773.ec. PMID 18332345
- [Background] Kalman LV, Tarleton JC, Percy AK, Aradhya S, Bale S, Barker SD, Bayrak-Toydemir P, Bridges C, Buller-Burckle AM, Das S, Iyer RK, Vo TD, Zvereff VV, Toji LH. Development of a genomic DNA reference material panel for Rett syndrome (MECP2-related disorders) genetic testing. J Mol Diagn. 2014 Mar;16(2):273-9. doi: 10.1016/j.jmoldx.2013.11.004. Epub 2014 Feb 7. PMID 24508304
- [Background] Leonard H, Ravikumara M, Baikie G, Naseem N, Ellaway C, Percy A, Abraham S, Geerts S, Lane J, Jones M, Bathgate K, Downs J; Telethon Institute for Child Health Research. Assessment and management of nutrition and growth in Rett syndrome. J Pediatr Gastroenterol Nutr. 2013 Oct;57(4):451-60. doi: 10.1097/MPG.0b013e31829e0b65. PMID 24084372
- [Background] Percy AK. Rett syndrome: exploring the autism link. Arch Neurol. 2011 Aug;68(8):985-9. doi: 10.1001/archneurol.2011.149. PMID 21825235
- [Background] Percy A. The American history of Rett syndrome. Pediatr Neurol. 2014 Jan;50(1):1-3. doi: 10.1016/j.pediatrneurol.2013.08.018. Epub 2013 Nov 5. No abstract available. PMID 24200039
- [Background] Neul JL, Glaze DG, Percy AK, Feyma T, Beisang A, Dinh T, Suter B, Anagnostou E, Snape M, Horrigan J, Jones NE. Improving Treatment Trial Outcomes for Rett Syndrome: The Development of Rett-specific Anchors for the Clinical Global Impression Scale. J Child Neurol. 2015 Nov;30(13):1743-8. doi: 10.1177/0883073815579707. Epub 2015 Apr 20. PMID 25895911
- [Result] Neul JL, Kaufmann WE, Glaze DG, Christodoulou J, Clarke AJ, Bahi-Buisson N, Leonard H, Bailey ME, Schanen NC, Zappella M, Renieri A, Huppke P, Percy AK; RettSearch Consortium. Rett syndrome: revised diagnostic criteria and nomenclature. Ann Neurol. 2010 Dec;68(6):944-50. doi: 10.1002/ana.22124. PMID 21154482
- [Result] Percy AK, Neul JL, Glaze DG, Motil KJ, Skinner SA, Khwaja O, Lee HS, Lane JB, Barrish JO, Annese F, McNair L, Graham J, Barnes K. Rett syndrome diagnostic criteria: lessons from the Natural History Study. Ann Neurol. 2010 Dec;68(6):951-5. doi: 10.1002/ana.22154. PMID 21104896
- [Result] Percy AK, Lee HS, Neul JL, Lane JB, Skinner SA, Geerts SP, Annese F, Graham J, McNair L, Motil KJ, Barrish JO, Glaze DG. Profiling scoliosis in Rett syndrome. Pediatr Res. 2010 Apr;67(4):435-9. doi: 10.1203/PDR.0b013e3181d0187f. PMID 20032810
- [Result] Glaze DG, Percy AK, Skinner S, Motil KJ, Neul JL, Barrish JO, Lane JB, Geerts SP, Annese F, Graham J, McNair L, Lee HS. Epilepsy and the natural history of Rett syndrome. Neurology. 2010 Mar 16;74(11):909-12. doi: 10.1212/WNL.0b013e3181d6b852. PMID 20231667
- [Result] Kirby RS, Lane JB, Childers J, Skinner SA, Annese F, Barrish JO, Glaze DG, Macleod P, Percy AK. Longevity in Rett syndrome: analysis of the North American Database. J Pediatr. 2010 Jan;156(1):135-138.e1. doi: 10.1016/j.jpeds.2009.07.015. PMID 19772971
- [Result] McCauley MD, Wang T, Mike E, Herrera J, Beavers DL, Huang TW, Ward CS, Skinner S, Percy AK, Glaze DG, Wehrens XH, Neul JL. Pathogenesis of lethal cardiac arrhythmias in Mecp2 mutant mice: implication for therapy in Rett syndrome. Sci Transl Med. 2011 Dec 14;3(113):113ra125. doi: 10.1126/scitranslmed.3002982. PMID 22174313
- [Result] Motil KJ, Caeg E, Barrish JO, Geerts S, Lane JB, Percy AK, Annese F, McNair L, Skinner SA, Lee HS, Neul JL, Glaze DG. Gastrointestinal and nutritional problems occur frequently throughout life in girls and women with Rett syndrome. J Pediatr Gastroenterol Nutr. 2012 Sep;55(3):292-8. doi: 10.1097/MPG.0b013e31824b6159. PMID 22331013
- [Result] Bebbington A, Downs J, Percy A, Pineda M, Zeev BB, Bahi-Buisson N, Leonard H. The phenotype associated with a large deletion on MECP2. Eur J Hum Genet. 2012 Sep;20(9):921-7. doi: 10.1038/ejhg.2012.34. Epub 2012 Apr 4. PMID 22473088
- [Result] Bebbington A, Percy A, Christodoulou J, Ravine D, Ho G, Jacoby P, Anderson A, Pineda M, Ben Zeev B, Bahi-Buisson N, Smeets E, Leonard H. Updating the profile of C-terminal MECP2 deletions in Rett syndrome. J Med Genet. 2010 Apr;47(4):242-8. doi: 10.1136/jmg.2009.072553. Epub 2009 Nov 12. PMID 19914908
- [Result] Tarquinio DC, Motil KJ, Hou W, Lee HS, Glaze DG, Skinner SA, Neul JL, Annese F, McNair L, Barrish JO, Geerts SP, Lane JB, Percy AK. Growth failure and outcome in Rett syndrome: specific growth references. Neurology. 2012 Oct 16;79(16):1653-61. doi: 10.1212/WNL.0b013e31826e9a70. Epub 2012 Oct 3. PMID 23035069
- [Result] Motil KJ, Barrish JO, Lane J, Geerts SP, Annese F, McNair L, Percy AK, Skinner SA, Neul JL, Glaze DG. Vitamin D deficiency is prevalent in girls and women with Rett syndrome. J Pediatr Gastroenterol Nutr. 2011 Nov;53(5):569-74. doi: 10.1097/MPG.0b013e3182267a66. PMID 21637127
- [Result] Lane JB, Lee HS, Smith LW, Cheng P, Percy AK, Glaze DG, Neul JL, Motil KJ, Barrish JO, Skinner SA, Annese F, McNair L, Graham J, Khwaja O, Barnes K, Krischer JP. Clinical severity and quality of life in children and adolescents with Rett syndrome. Neurology. 2011 Nov 15;77(20):1812-8. doi: 10.1212/WNL.0b013e3182377dd2. Epub 2011 Oct 19. PMID 22013176
- [Result] Chapleau CA, Lane J, Kirwin SM, Schanen C, Vinette KM, Stubbolo D, MacLeod P, Glaze DG, Motil KJ, Neul JL, Skinner SA, Kaufmann WE, Percy AK. Detection of rarely identified multiple mutations in MECP2 gene do not contribute to enhanced severity in Rett syndrome. Am J Med Genet A. 2013 Jul;161A(7):1638-46. doi: 10.1002/ajmg.a.35979. Epub 2013 May 21. PMID 23696494
- [Result] Cuddapah VA, Pillai RB, Shekar KV, Lane JB, Motil KJ, Skinner SA, Tarquinio DC, Glaze DG, McGwin G, Kaufmann WE, Percy AK, Neul JL, Olsen ML. Methyl-CpG-binding protein 2 (MECP2) mutation type is associated with disease severity in Rett syndrome. J Med Genet. 2014 Mar;51(3):152-8. doi: 10.1136/jmedgenet-2013-102113. Epub 2014 Jan 7. PMID 24399845
- [Result] Neul JL, Lane JB, Lee HS, Geerts S, Barrish JO, Annese F, Baggett LM, Barnes K, Skinner SA, Motil KJ, Glaze DG, Kaufmann WE, Percy AK. Developmental delay in Rett syndrome: data from the natural history study. J Neurodev Disord. 2014;6(1):20. doi: 10.1186/1866-1955-6-20. Epub 2014 Jul 22. PMID 25071871
- [Result] Killian JT, Lane JB, Cutter GR, Skinner SA, Kaufmann WE, Tarquinio DC, Glaze DG, Motil KJ, Neul JL, Percy AK. Pubertal development in Rett syndrome deviates from typical females. Pediatr Neurol. 2014 Dec;51(6):769-75. doi: 10.1016/j.pediatrneurol.2014.08.013. Epub 2014 Aug 29. PMID 25283752
- [Result] Tarquinio DC, Hou W, Neul JL, Lane JB, Barnes KV, O'Leary HM, Bruck NM, Kaufmann WE, Motil KJ, Glaze DG, Skinner SA, Annese F, Baggett L, Barrish JO, Geerts SP, Percy AK. Age of diagnosis in Rett syndrome: patterns of recognition among diagnosticians and risk factors for late diagnosis. Pediatr Neurol. 2015 Jun;52(6):585-91.e2. doi: 10.1016/j.pediatrneurol.2015.02.007. Epub 2015 Feb 16. PMID 25801175
- [Derived] Buchanan CB, Stallworth JL, Joy AE, Dixon RE, Scott AE, Beisang AA, Benke TA, Glaze DG, Haas RH, Heydemann PT, Jones MD, Lane JB, Lieberman DN, Marsh ED, Neul JL, Peters SU, Ryther RC, Skinner SA, Standridge SM, Kaufmann WE, Percy AK. Anxiety-like behavior and anxiolytic treatment in the Rett syndrome natural history study. J Neurodev Disord. 2022 May 14;14(1):31. doi: 10.1186/s11689-022-09432-2. PMID 35568815
- See also: Click here for the International Rett Syndrome Foundation website — http://www.rettsyndrome.org/